CLINICAL TRIAL: NCT05036642
Title: Effects of Post-Stroke Upper Extremity Assistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Allison Okamura, Professor of Mechanical Engineering, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-61540; SNI-BI1-02 (Other Grant/Funding Number: Stanford Neurosciences Institute)
Record Dates: First submitted 2021-08-31; First posted 2021-09-05 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Arm Weakness as a Consequence of Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Stroke Survivors (Experimental): Stroke survivors with upper extremity motor impairments
  Interventions: Device: Compliant Passive Arm Support

INTERVENTIONS:
Device: Compliant Passive Arm Support — The device is a mechanical device that consists of two linkages, elastic bands, a commercial posture brace, and a hook-and-loop fastener. The design of the device, with several compliant elements, ensures that one device fits many without joint alignment concerns. No motors or other actuators add energy into the system, meaning that it is stable.

SUMMARY:
The purpose of this study is to quantify the improvement of post- stroke individuals' ability to move their arms during and after robot assisted therapy.

While researchers know that robot assisted therapies improve motor performance over the course of weeks, they do not know how motor performance is affected over the course of minutes or hours. A better understanding of how robot assisted therapies affect motor performance on short time scales may help us to prescribe more effective therapy doses to maximize motor recovery after neurological injury.

The study will allow us to obtain a detailed understanding of the performance of the device as described above.

ELIGIBILITY:
Inclusion Criteria:

* greater than 6 months post-stroke
* passive abduction to 90 degrees at shoulder
* reduced active (retro)flexion/extension at shoulder when abducted at 90 degrees
* reduced active flexion/extension at elbow

Exclusion Criteria:

* unable to give informed consent
* unable to comprehend and follow instructions
* have a condition (other than stroke) affecting sensorimotor function
* show evidence of unilateral spatial neglect
* unable to sit in a chair without armrests for 2 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Okamura, Principal Investigator — Stanford University
Locations (1):
- Stanford University CHARM Lab, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sukal TM, Ellis MD, Dewald JP. Shoulder abduction-induced reductions in reaching work area following hemiparetic stroke: neuroscientific implications. Exp Brain Res. 2007 Nov;183(2):215-23. doi: 10.1007/s00221-007-1029-6. Epub 2007 Jul 20. PMID 17634933

RESULTS

PARTICIPANT FLOW:
Groups:
- Pilot Phase: Pilot testing by stroke survivors with upper extremity motor impairments use a Compliant Passive Arm Support. The device is a mechanical device that consists of two linkages, elastic bands, a commercial posture brace, and a hook-and-loop fastener. The design of the device, with several compliant elements, ensures that one device fits many without joint alignment concerns. No motors or other actuators add energy into the system, meaning that it is stable.
- Evaluation Phase: Stroke survivors with upper extremity motor impairments use a Compliant Passive Arm Support. The device is a mechanical device that consists of two linkages, elastic bands, a commercial posture brace, and a hook-and-loop fastener. The design of the device, with several compliant elements, ensures that one device fits many without joint alignment concerns. No motors or other actuators add energy into the system, meaning that it is stable.
Period: Pilot Phase
Arm/Group | Pilot Phase | Evaluation Phase
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0
Period: Evaluation Phase
Arm/Group | Pilot Phase | Evaluation Phase
Started | 0 | 11
Completed | 0 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pilot Phase: Pilot testing by stroke survivors with upper extremity motor impairments use a Compliant Passive Arm Support.
- Evaluation Phase: Stroke survivors with upper extremity motor impairments use a Compliant Passive Arm Support.
- Total: Total of all reporting groups
Arm/Group | Pilot Phase | Evaluation Phase | Total
Number analyzed (Participants) | 1 | 11 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 4 | 4
  >=65 years | 1 | 7 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 1 | 8 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 11 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 5 | 6
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 11 | 12

OUTCOME MEASURES:

1. Primary Outcome: Wolf Motor Function Test - Change in Functional Score by Task (WMFT)
Description: Change reported as number of tasks where participants on average had increased functionality, no change, or decreased functionality. Lower functional scores are indicative of lower functional levels. The WMFT consists of 17 tasks: Forearm to table (side), Forearm to box (side), Extend elbow (to the side), Extend elbow (to the side) - with weight, Hand to table (front), Hand to box (front), Weight to box, Reach and retrieve, Lift can, Lift pencil, Lift paper clip, Stack checkers, Flip cards, Grip Strength, Turning key In lock, Fold towel, and Lift basket. Fifteen tasks were assessed for this outcome: task 7 (Weight to box) is reported in a separate analysis; task 14 (Grip strength) was excluded due to an inability to acquire the necessary equipment.
Time Frame: Assessed at baseline (without the device) and after approximately 30 minutes of use with the device.
Population: Data for this outcome were collected from participants in the Evaluation phase only.
Measure: Count of Units; unit: Tasks
Units Other Than Participants: Tasks
Arm/Group | Evaluation Phase
Number analyzed (Participants) | 11
Number analyzed (Tasks) | 15
Tasks
  Increase functionality | 7
  No change | 3
  Decreased functionality | 5

2. Primary Outcome: Wolf Motor Function Test - Change in Completion Time by Task
Description: Change reported as number of tasks which participants on average performed with increased time, no change, or decreased time. If a participant was unable to complete the task, a time score of 120+ seconds was assigned and converted to 121 for calculation purposes. The WMFT consists of 17 tasks: Forearm to table (side), Forearm to box (side), Extend elbow (to the side), Extend elbow (to the side) - with weight, Hand to table (front), Hand to box (front), Weight to box, Reach and retrieve, Lift can, Lift pencil, Lift paper clip, Stack checkers, Flip cards, Grip Strength, Turning key In lock, Fold towel, and Lift basket. Fifteen tasks were assessed for this outcome: task 7 (Weight to box) is reported in a separate analysis; task 14 (Grip strength) was excluded due to an inability to acquire the necessary equipment.
Time Frame: Assessed at baseline (without the device) and after approximately 30 minutes of use with the device.
Population: Data for this outcome were collected from participants in the Evaluation phase only.
Measure: Count of Units; unit: Tasks
Units Other Than Participants: Tasks
Arm/Group | Evaluation Phase
Number analyzed (Participants) | 11
Number analyzed (Tasks) | 15
Tasks
  Increased time | 3
  No change | 0
  Decreased time | 12

3. Primary Outcome: Wolf Motor Function Test - Weight Lifted
Description: Weight lifted (carried) in task 7 of the WMFT: Weight to box. In this assessment, the participant is seated and lifts weight to a box centered on a table in front of them, while keeping his/her back against the chair.
Time Frame: Assessed at baseline (without the device) and after approximately 5 minutes of use with the device.
Population: Data for this outcome were collected from participants in the Evaluation phase only.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Evaluation Phase
Number analyzed (Participants) | 11
pounds
  No Device | 4.6 (4.8)
  With Device | 6.1 (4.8)

4. Primary Outcome: Percentage of Successful Motions
Description: Participants are instructed to individually flex and extend the elbow and shoulder to trace the largest possible circle that they can reach while keeping the hand and elbow raised to the height of the shoulder while the motion of the arm is tracked with motion capture. The participant was asked to perform 6 motions (3 clockwise and 3 counterclockwise in randomized order). This protocol was originally developed by Sukal et al (2007); to asses post-stroke motor abilities. Successful motion is defined as motion where any part of the arm is within 20cm of shoulder level. The percentage of motion in which successful motion occurred over the total motion was reported.
Time Frame: Assessed at baseline (without the device) and after approximately 30 minutes of use with the device.
Population: Data for this outcome were collected from participants in the Evaluation phase only.
Measure: Mean (Standard Deviation); unit: percentage of motions
Units Other Than Participants: Motions
Arm/Group | Evaluation Phase
Number analyzed (Participants) | 11
Number analyzed (Motions) | 6
percentage of motions
  No device | 57.5 (42.28)
  With device | 69.84 (45.07)
Statistical Analysis 1: Comparison: Evaluation Phase; Difference in measurements from 'no device' (baseline) to 'with device.'; Test type: Other; p = 0.02, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Reachable Workspace - Mean Distance From Trunk, Successful Motions
Description: Participants are instructed to individually flex and extend the elbow and shoulder to trace the largest possible circle that they can reach while keeping the hand and elbow raised to the height of the shoulder while the motion of the arm is tracked with motion capture. This protocol was originally developed by Sukal et al (2007); to asses post-stroke motor abilities. Successful motion is defined as motion where any part of the arm is within 20cm of shoulder level. The distance from the wrist to the trunk was reported for successful motion. Distance closer to the trunk indicates greater ability to correctly perform the task. Negative numbers would indicate the arm was below the trunk; positive numbers would indicate the arm was above the trunk.
Time Frame: Assessed at baseline (without the device) and after approximately 30 minutes of use with the device.
Population: Data for this outcome were collected from participants in the Evaluation phase only.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Evaluation Phase
Number analyzed (Participants) | 11
meters
  No device | -0.07 (0.07)
  With device | -0.05 (0.07)
Statistical Analysis 1: Comparison: Evaluation Phase; Difference in measurements from 'no device' (baseline) to 'with device.'; Test type: Other; p = 0.01, ANOVA

6. Primary Outcome: Reachable Workspace - Area, Successful Motions
Description: Participants will be instructed to individually flex and extend the elbow and shoulder to trace the largest possible circle that they can reach while keeping the hand and elbow raised to the height of the shoulder while the motion of the arm is tracked with motion capture. This protocol was originally developed by Sukal et al (2007); to asses post-stroke motor abilities. A larger workspace area indicates fewer upper extremity motor impairments.
Time Frame: Assessed at baseline (without the device) and after approximately 30 minutes of use with the device.
Population: Data for this outcome were collected from participants in the Evaluation phase only.
Measure: Mean (Standard Deviation); unit: m^2
Arm/Group | Evaluation Phase
Number analyzed (Participants) | 11
m^2
  No device | 0.078 (0.084)
  With device | 0.082 (0.073)
Statistical Analysis 1: Comparison: Evaluation Phase; Difference in measurements from 'no device' (baseline) to 'with device.'; Test type: Other; p = 0.48, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Reachable Workspace - Mean Distance From Trunk, All Motions
Description: Participants are instructed to individually flex and extend the elbow and shoulder to trace the largest possible circle that they can reach while keeping the hand and elbow raised to the height of the shoulder while the motion of the arm is tracked with motion capture. This protocol was originally developed by Sukal et al (2007); to asses post-stroke motor abilities. The distance from the wrist to the trunk was reported for all motion. Distance closer to the trunk indicates greater ability to correctly perform the task. Negative numbers would indicate the arm was below the trunk; positive numbers would indicate the arm was above the trunk.
Time Frame: Assessed at baseline (without the device) and after approximately 60 minutes of use with the device.
Population: Data for this outcome were collected from participants in the Evaluation phase only.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Evaluation Phase
Number analyzed (Participants) | 11
meters
  No device | -0.14 (0.12)
  With device | -0.12 (0.12)

8. Secondary Outcome: Participant Satisfaction Survey
Description: Closing survey of participants satisfaction with the device (impact, comfort, and responsiveness). Participants rated the experience as very positive, positive, neutral, negative, or very negative.
Time Frame: After study procedures have been performed, on day 2 (up to 5 minutes to complete survey)
Population: Data for this outcome were collected from participants in the Evaluation phase only. Participants who completed the survey are included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Very Positive; Positive; Neutral; Negative; Very Negative: Stroke survivors with upper extremity motor impairments use a Compliant Passive Arm Support.
Arm/Group | Very Positive | Positive | Neutral | Negative | Very Negative
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Participants
  Impact | 3 | 4 | 1 | 1 | 1
  Comfort | 4 | 1 | 0 | 5 | 0
  Responsiveness | 2 | 6 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Pilot Phase | Evaluation Phase
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/11
Other Adverse Events (participants affected / at risk) | 0/1 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT05036642/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT05036642/SAP_001.pdf